CLINICAL TRIAL: NCT03160170
Title: Intraoperative Efficacy of Suction Enabled Retraction Device in Lumbar Spine Surgery
Brief Title: Efficacy of Suction Enabled Retraction Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources no longer available
Sponsor: University of Miami (Other)
Collaborators: Ludwig Medical Corporation (Unknown)
Responsible Party: Principal Investigator, Ian Cote, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20161061
Record Dates: First submitted 2017-05-15; First posted 2017-05-19 (Actual); Results first posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-04

CONDITIONS: Surgical Blood Loss; Spinal Surgery
Keywords: open lumbar spine surgery; operative time and efficiency; Suction-Integrated Surgical Tissue Elevator and Retractor
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Use of Cobb device (Experimental): Use of SISTER device during surgery
  Interventions: Device: SISTER device
- Control (No Intervention): Standard exposure technique and instruments will be used during surgery

INTERVENTIONS:
Device: SISTER device — Use of the Suction-Integrated Surgical Tissue Elevator & Retractor (SISTER) device during surgery
  Other Names: Cobb
  Arms: Use of Cobb device

SUMMARY:
This is a prospective randomized controlled trial of the Suction-Integrated Surgical Tissue

Elevator & Retractor [SISTER] device to assess:

* Effects on operative time and efficiency of exposure in open lumbar spine cases.
* Effect on total blood loss during the exposure part of the operation.
* Rate of clogging of suction device.

DETAILED DESCRIPTION:
The device, Suction-Integrated Surgical Tissue Elevator & Retractor [SISTER], is shaped like a Cobb elevator but also has a hollow core allowing suction tubing to be connected. Thus, a single hand can be used to retract and suction at the same time while the other hand separates soft tissue from the bones with electrocautery. This set up which is proposed to be more efficient will be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Patients undergoing lumbar one to sacral one open instrumentation
* Surgery performed by the Departments of Neurological Surgery and Orthopedics at the University of MIami Miller School of Medicine

Exclusion Criteria:

* Less than 22 years old
* Procedure does not involve instrumentation
* Prior lumbar spine surgery involving more than one level
* BMI less than 20 or greater than 35
* Known bleeding conditions ( ex. Factor V Leiden, Von Willebrand)
* Routinely taking anticoagulation medicine (ex. aspirin 325 mg/day, Plavix)
* Operative cases where a single surgeon performs both sides of exposure
* Pregnant women
* Prisoners
* Adults unable to consent

Ages: 22 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Cõté, MD, Principal Investigator — University of Miami
Locations (1):
- Jackson Memorial Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Use of Cobb Device | Control
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Use of Cobb Device | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (11.8) | 71.1 (7.4) | 68.2 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 8 | 6 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Estimated Blood Loss
Description: Amount of blood loss from incision time to screw placement
Time Frame: 1.5 hours
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Use of Cobb Device | Control
Number analyzed (Participants) | 10 | 10
ml | 364.0 (363.1) | 356.0 (256.5)
Statistical Analysis 1: Comparison: Use of Cobb Device vs Control; Test type: Superiority; p = 0.96, t-test, 2 sided

2. Secondary Outcome: Time of Exposure
Description: Length of operation in minutes
Time Frame: 1.5 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Use of Cobb Device | Control
Number analyzed (Participants) | 10 | 10
minutes | 38.2 (9.0) | 69.7 (56.1)
Statistical Analysis 1: Comparison: Use of Cobb Device vs Control; Test type: Superiority; p = 0.11, t-test, 2 sided

3. Secondary Outcome: Rate of Clogging
Description: Average number of times the suction tip of the device had to be unclogged
Time Frame: 1.5 hours
Measure: Mean (Standard Deviation); unit: tip clogs
Arm/Group | Use of Cobb Device | Control
Number analyzed (Participants) | 10 | 10
tip clogs | 10.1 (4.9) | 4.9 (6.0)
Statistical Analysis 1: Comparison: Use of Cobb Device vs Control; Test type: Superiority; p = 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1.5 hours
Arm/Group | Use of Cobb Device | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/70/NCT03160170/Prot_SAP_000.pdf